CLINICAL TRIAL: NCT01494077
Title: Accuracy of Dilution of EUS-FNA Pancreatic Cyst Fluid for CEA Measurement
Brief Title: Accuracy of Dilution of EUS-FNA Pancreatic Cyst Fluid for Carcinoembryonic Antigen (CEA) Measurement
Status: Completed | Type: Observational
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Kenneth J. Chang, Professor of Clinical Medicine, University of California, Irvine
Other Study IDs: HS#2011-8161
Record Dates: First submitted 2011-12-02; First posted 2011-12-16 (Estimated); Last update posted 2014-12-12 (Estimated); Status verified 2014-12

CONDITIONS: Pancreatic Cyst
Keywords: Pancreatic Cyst Fluid; Dilution; Carcinoembryonic Antigen (CEA)
MeSH Terms: conditions — Pancreatic Cyst

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- EUS-FNA of Pancreatic Cyst: Patients who have a pancreatic cyst requiring standard of care EUS-FNA that yields 2.25 ML (or greater) of fluid will be included in the study.
  Interventions: Other: Laboratory processing for results

INTERVENTIONS:
Other: Laboratory processing for results — There is no intervention. Extra fluid that is normally discarded will be processed.

SUMMARY:
The purpose of this research project is to determine if pancreatic cyst fluid can be diluted and provide an accurate Carcinoembryonic Antigen (CEA) level. The investigators hypothesis is that pancreatic cyst fluid obtained by EUS-FNA can be diluted effectively and accurately for the measurement of CEA levels.

DETAILED DESCRIPTION:
Potential subjects will be identified based on the indication of a pancreatic cyst requiring EUS-FNA. The procedure will be performed as usual per standard protocol with EUS-FNA of the cyst. Once the fluid is aspirated, it will be measured and if the fluid volume is 2.25 mL or greater than the patient will be included in the study.

A micropipette will be used to ensure exact volumes are measured. The first 1 mL of cystic fluid will be sent to the lab for regular CEA analysis, per standard protocol. The remaining fluid, which would usually be discarded, will then be used for the study. The micropipette will be used to mix 0.75 mL of cyst fluid with 0.25 mL of normal saline (designated sample #2). Next, 0.5 mL of cyst fluid will be mixed with 0.5 mL of normal saline for the next study sample (designated sample #3). These two study samples will be sent to the lab separately using de-identified information, and these values will not be part of the patient's medical record and will not affect clinical management or decision-making. The study samples will be given a unique identifier that will not have any patient identification. The unique identifier will allow the study researchers to link the values to the correct patient by using a password protected program that cannot be accessed by the public.

This study will not require any additional patient participation, and will not impact the length of the procedure. The only additional time will be from the study researchers and the EUS technologists diluting the samples, which will not affect the procedure time itself. If a single patient has more than one cyst, each cyst can be included in the study separately. No additional photographs, videos or data other than the standard data for the procedure will be produced.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for EUS-FNA of a pancreatic cyst
* Cyst must yield 2.25ml (or greater) of fluid

Exclusion Criteria:

* Cysts yielding less than 2.25ml of fluid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are already scheduled for EUS-FNA of a pancreatic cyst at the H.H. Chao Comprehensive Digestive Disease Center at UC Irvine Medical Center. The procedure will be performed as usual per standard of care protocol with EUS-FNA of the cyst. Once the fluid is aspirated, it will be measured and if the fluid volume is 2.25 mL or greater than the patient will be included in the study.
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2011-04; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Accuracy of diluted CEA level | Pancreatic fluid is aspirated once during the procedure.
  The primary aim of this study is to determine if pancreatic cyst fluid can be diluted and provide an accurate CEA level.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth J. Chang, MD, Principal Investigator — University of California, Irvine
Locations (1):
- H. H. Chao Comprehensive Digestive Disease Center, Orange, California, United States